CLINICAL TRIAL: NCT00005064
Title: Phase I Study of PS-341 in Acute Myeloid Leukemias, Myelodysplastic Syndromes and Chronic Myeloid Leukemia in Blast Phase
Brief Title: PS-341 in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Chronic Myeloid Leukemia in Blast Phase, or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02322; DM 99-245; U01CA062461 (NIH); CDR0000067668 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2004-02-02 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Acute Promyelocytic Leukemia (M3); Blastic Phase Chronic Myelogenous Leukemia; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive PS-341 IV bolus twice weekly for 4 weeks followed by 2 weeks of rest. Treatment continues for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Phase I trial to study the effectiveness of PS-341 in treating patients who have refractory or relapsed acute myeloid leukemia, acute lymphoblastic leukemia, chronic myeloid leukemia in blast phase, or myelodysplastic syndrome. PS-341 may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of PS-341 in patients with refractory or relapsed acute myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, or chronic myeloid leukemia in blast phase.

II. Assess the plasma pharmacology of this drug, its ability to inhibit proteasome function and to accelerate apoptosis in circulating blasts in this patient population.

III. Assess the antileukemic effects of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive PS-341 IV bolus twice weekly for 4 weeks followed by 2 weeks of rest. Treatment continues for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 2 patients receive escalating doses of PS-341 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose level associated with toxicity probability closest to 0.2 after 30 patients are treated.

ELIGIBILITY:
Inclusion Criteria:

* AML, ALL, or high-risk MDS (R-AEB or RAEB-t) that has:

  * Not responded (no CR) to initial induction chemotherapy, or
  * Recurred after an initial CR of < 1 year, or
  * Recurred after an initial CR of > 1 year and failed to respond to an initial re-induction attempt, or
  * Recurred more than once, OR
* Chronic myeloid leukemia in myeloid blast phase

  * Patients with CML blast phase may receive PS-341 as their first therapy for blast phase or after failing other treatments for blast phase
* Patients with refractory or relapsed acute promyelocytic leukemia are eligible provided they have failed an ATRA-containing regimen
* Patients who are likely to benefit from allogeneic bone marrow transplantation (i.e., age < 60 years of physiological age with histocompatible donor) should be excluded from this study unless such therapy is not feasible
* ECOG performance status =< 52 (Karnofsky >= 50%)
* Total bilirubin < 1.6 mg/ml
* ALT or AST =< 2.5 times the institutional upper limit of normal
* Creatinine < 1.6 mg/ml or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy; use of hydroxyurea on patients with rapidly proliferative disease (i.e., absolute peripheral blood blast count >= 5 x 10^9/L, and increasing by >= 1 x 10^9/L/24 hrs) is allowed up to 24 hours prior to the start of therapy with PS-341
* The effects of PS-341 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Because the potential risk of toxicity in nursing infants secondary to PS-341 treatment of the mother is unknown but may be harmful, breastfeeding should be discontinued if the mother is treated with PS-341
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients undergoing therapy with other investigational agents
* Patients with known brain metastases or CNS disease should be excluded from this clinical trail because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other toxicities
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia
* HIV-positive patients receiving, anti-retroviral thearpy (HAART) are excluded from the study because of possible pharmacokinetic interactions; appropriate studies will be undertaken in patients receiving, HAART therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-02; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of greater or equal grade 3 toxicity | 35 days
  Graded using the NCI CTC version 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States